CLINICAL TRIAL: NCT05993650
Title: Inspiratory Muscle Training in Individuals With Chronic Venous Disease : A Randomized Controlled Study
Brief Title: Inspiratory Muscle Training in Chronic Venous Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Özlem Çınar Özdemir, Assoc. prof, Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IMT in Venous Diseases
Record Dates: First submitted 2023-07-31; First posted 2023-08-15 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Chronic Venous Insufficiency
Keywords: chronic venous insufficiency; maximal respiratory pressures; respiratory function tests; exercise capacity; edema; pain; quality of life
MeSH Terms: conditions — Edema; Pain

STUDY DESIGN:
Intervention Model Description: Assessment
Who Masked: Participant
Masking Description: Single-blind study; the patients will not be informed about training group or control group and they will be evaluated and trained at different places and times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): The individuals in the training group will be performed inspiratory muscle training using an inspiratory muscle training device (PowerBreathe®) at 30-50% of the maximal inspiratory pressure.
  Interventions: Other: Inspiratuar Muscle Training Group
- Control Group (Sham Comparator): Individuals in this group will be given thoracic expansion exercises and patient education.
  Interventions: Other: Thoracic Expansion Exercise Group

INTERVENTIONS:
Other: Inspiratuar Muscle Training Group — Inspiratory muscle training will be done for 15 minutes/session, 2 times/day, or 30 minutes/day if tolerated, 5-7 days/week (one under supervision and others at home), for a total of 6 weeks. Applications made at home will be followed with a diary. Inspiratory muscle training will be performed using an inspiratory muscle training device (PowerBreathe®) working with the threshold loading principle.In the first week of the training, 30-50% of the maximal inspiratory pressure (MIP) measured in the initial evaluation of the individual will be adjusted according to the patient's tolerance, and inspiratory muscle training will be performed. Respiratory muscle strength measurement will be repeated every week in the individuals in the training group. 30-50% of the new MIP value obtained will be calculated and adjusted by calculating the new training workload for the application of inspiratory muscle training in the following weeks
  Other Names: Inspiratuar Muscle Training
  Arms: Training Group
Other: Thoracic Expansion Exercise Group — Individuals in this group will be given thoracic expansion exercises and patient education. Thoracic expansion exercises will be applied to individuals in an upright sitting position. In this position, individuals will place their hands on their lower ribs and then perform the cycle of "inhale a deep breathing + holding the deep breath for 3 seconds + slowly exhale all the breath" 3 times in a row. After this cycle, individuals will be asked to rest by taking 3-4 calm breaths. Immediately after, the individual will be asked to repeat the same cycle and repeat the cycle with calm breaths and rest until it reaches 10 repetitions. The individual will do this session 4 times a day. Individuals will do the first session of breathing exercises under supervision. In this way, incorrect exercise will be prevented. Other breathing exercise sessions will be done by individuals as a home program every day and 4 sessions a day during 6 weeks.
  Arms: Control Group

SUMMARY:
There is insufficient evidence of inspiratory muscle training on venous function, clinical severity, symptoms and functional capacity and quality of life in CVI patients. Therefore, in the study, the investigators aimed to determine the effectiveness of inspiratory muscle training in individuals with chronic venous insufficiency.

DETAILED DESCRIPTION:
Chronic venous insufficiency (CVI) is defined as a very common condition that affects the venous system in the lower extremities, including various pathologies and subjective symptoms such as pain, cramps, restlessness in the legs, edema, itching and skin changes. CVI is a disease that develops due to venous hypertension in the lower extremities, resulting in impaired turbulent flow fields, venous distention, free radical formation and inflammation. In addition to being a cosmetic problem, symptoms such as pain, itching, burning, tingling, night cramps, edema, skin changes and venous ulcers in chronic cases can be seen. It is seen between 5-30% in the adult population. CVI affects 40% of the general population. Because of its high prevalence, chronic venous diseases are a common condition that causes major socioeconomic impacts. According to the studies; it has been observed that 32% of women and 40% of men have varicose veins, and any type of venous disease affects 40-50% of men and 50-55% of.

The main clinical features of CVI are dilated veins, edema, leg pain, muscle cramps, and cutaneous changes in the leg. Edema begins in the perimalleolar region and ascendes up the leg. Leg restlessness is often described as heaviness or pain after prolonged standing and is relieved by leg elevation. This discomfort is caused by increased intracompartmental and subcutaneous volume and pressure. Venous valves and venous pump are the two major determinants of venous flow. Venous valves play a role in directing the flow from the superficial system to the deep system and in its progression from the proximal veins to the distal veins.

Venous function is reflected in venous return, venous resistance, and its effects on cardiac output. Venous filling time is a parameter of venous function and is shortened as a result of valve insufficiency, vessel wall enlargement and inability of muscle pumps to work actively. The calf muscles compress the deep intramuscular veins, diverting blood flow from the veins to the heart. This mechanism depends on talocrural mobility and the force of contraction of the calf muscles. However, muscle pump dysfunction is not limited to the calf, but also includes inspiratory muscle dysfunction, such as when the diaphragm allows greater blood flow to the heart from the lower extremities, creating a suction effect on the inferior vena cava during inspiration and expiration. It has been shown that the respiratory cycle affects the increase of deep inspiration and the flow rate of the femoral vein and venous return in healthy individuals. When inspiratory muscle strength is insufficient, blood flow in the leg veins will decrease, increasing vascular resistance and thus systemic refill can be reduced. Increasing the muscle strength of inspiration with inspiratory muscle training is considered to increase venous return and improve symptoms of CVI, including pain and edema. However, there is insufficient evidence of inspiratory muscle training on venous function, clinical severity, symptoms and functional capacity and quality of life in CVI patients. Therefore, in the study, the investigators aimed to determine the effectiveness of inspiratory muscle training in individuals with chronic venous insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with CVI
* Being between C1-C5 according to the 'Clinical, Etiologic, Anatomic, Pathophysiologic' (CEAP) scale,
* To accept to participate in the study,

Exclusion Criteria:

* Arterial diseases,
* Presence of advanced cardiorespiratory diseases,
* Having orthopedic and neurological disorders that may affect walking,
* Presence of acute ulcer (< 3 months) and diabetic ulcers,
* Being pregnant.
* Having a history of deep vein thrombosis,
* Having undergone venous system surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Maximal inspiratory pressure (MIP) | After 6-week training
  The MIP which shows respiratory muscle strength will be evaluated using a portable mouth pressure measuring device based on American Thoracic Society and European Respiratory Society criteria.

SECONDARY OUTCOMES:
Maximal expiratory pressure (MEP) | After 6-week training
  The MEP which shows respiratory muscle strength will be evaluated using a portable mouth pressure measuring device based on American Thoracic Society and European Respiratory Society criteria.
Forced vital capacity (FVC) | After 6-week training.
  Pulmonary function (Forced vital capacity (FVC)) will be evaluated with a spirometer. In the study, measurements will be made using the Cosmed Omnia microQuark 1.5 (Cosmed, Rome, Italy) device. Considering that dizziness may occur during forced expiration, measurements will be made while individuals are in a sitting position. While participants are sitting in a comfortable position in a chair with a backrest, nose clip will be attached and they will be asked to bite the mouthpieces with their teeth and close their lips in a way that does not allow air to escape. The tests will be performed at least 3 times by the participants and care will be taken to ensure that the expiration time is at least 6 seconds and the plateau time is 1 second. Due to the device software that records all three data, it saves the average of the two best data and processes it as a value.
Forced expiratory volume in the first second (FEV1) | After 6-week training.
  Pulmonary function (Forced expiratory volume in the first second (FEV1)) will be evaluated with a spirometer.
FEV1 / FVC | After 6-week training.
  Pulmonary function (FEV1 / FVC) will be evaluated with a spirometer.
Flow rate 25-75% of forced expiratory volume (FEF 25-75%) | After 6-week training.
  Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) will be evaluated with a spirometer.
Peak flow rate (PEF) | After 6-week training.
  Pulmonary function (Peak flow rate (PEF)) will be evaluated with a spirometer.
Aerobic capacity assessment | After 6-week training.
  The six-minute walk test (6-MWT) will be performed according to the criteria of the American Thoracic Society for the evaluation of aerobic capacity.
Lower extremity strength | After 6-week training.
  To determine lower extremity strength and functional mobility, the 30-second Sit-Up Test will be used in the chair
Edema assessment | After 6-week training.
  It is planned to evaluate the edema in the lower extremity by measuring the circumference with a tape measure. Both legs will be recorded separately and the difference will be calculated. A bendable, non-elastic, 7 mm wide standard tape measure with an accuracy of 0.1 cm will be used for circumference measurements. The "0" (zero) end of the tape measure will be wrapped around the area to be measured, with the "0" (zero) end in the left hand and the other end in the right hand, and the number above the "0" (zero) point will be noted
Quality of life assessment | After 6-week training.
  Quality of life will be evaluated using Chronic Venous Disease Quality of Life Questionnaire (CIVIQ-20).CIVIQ-20 is a quality of life survey that contains 20 questions and is specific for Chronic Venous Insufficiency, encompassing four quality of life domains: physical, psychological and social impairment and the severity of pain. There is a 5-point answer rating in each question, according to which higher scores indicate more severe impairment. There is a score varying from 0 to 100 in the CIVIQ-20 where the higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Çinar Özdemir, Study Director — Izmir Democracy University; Gülşah BARĞI, Principal Investigator — Izmir Democracy University; Cemre GÖRÜNMEZOĞLU, MSc, Principal Investigator — Izmir Democracy University; Dündar Özalp KARABAY, Principal Investigator — Dokuz Eylul University
Locations (1):
- Izmir Democracy University, Izmir, Karabağlar/İZMİR, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] OZDEMIR, Özlem Çınar; BAKAR, Yeşim; SÜRMELI, Mahmut. Kronik Venöz Yetmezlikte Ağrı, Yaşam Kalitesi Ve Depresyon Arasındaki İlişkinin İncelenmesi. Konuralp Medical Journal/Konuralp Tip Dergisi, 2017, 9.2.
- [Background] Aydin G, Yeldan I, Akgul A, Ipek G. Effects of inspiratory muscle training versus calf muscle training on quality of life, pain, venous function and activity in patients with chronic venous insufficiency. J Vasc Surg Venous Lymphat Disord. 2022 Sep;10(5):1137-1146. doi: 10.1016/j.jvsv.2022.04.012. Epub 2022 Jun 14. PMID 35710091
- [Background] Kwon OY, Jung DY, Kim Y, Cho SH, Yi CH. Effects of ankle exercise combined with deep breathing on blood flow velocity in the femoral vein. Aust J Physiother. 2003;49(4):253-8. doi: 10.1016/s0004-9514(14)60141-0. PMID 14632624
- [Background] Ozdemir OC, Tonga E, Tekindal A, Bakar Y. Cross-cultural adaptation, reliability and validity of the Turkish version of the Chronic Venous Disease Quality of Life Questionnaire (CIVIQ-20). Springerplus. 2016 Mar 31;5:381. doi: 10.1186/s40064-016-2039-2. eCollection 2016. PMID 27066388